CLINICAL TRIAL: NCT01347177
Title: A Single-centre Randomised Controlled Clinical Trial of Zirconia-based Versus Metal-based Adhesive Bridges for Replacing 2 Missing Teeth or Less in Adults.
Brief Title: Clinical Trial of Zirconia and Metal Adhesive Bridges
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100298307
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2011-01

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zirconia-based adhesive bridges (Experimental): Patients in this group will be treated with the employment of zirconia-based adhesive bridges to replace the missing tooth/teeth.
  Interventions: Procedure: Zirconia-based adhesive bridge
- Metal-based adhesive bridges (Experimental): Patients in this group will be treated with the employment of metal-based adhesive bridges.
  Interventions: Procedure: Metal-based adhesive bridge

INTERVENTIONS:
Procedure: Zirconia-based adhesive bridge — Zirconia-based adhesive bridge will be used to replace the missing tooth/teeth.
  Arms: Zirconia-based adhesive bridges
Procedure: Metal-based adhesive bridge — The metal-based adhesive bridge will be used to replace the missing tooth/teeth.
  Arms: Metal-based adhesive bridges

SUMMARY:
Adhesive bridges are becoming popular in patients with congenitally missing teeth and these are type of bridges that can be done with only minimal or with no preparation to replace the missing tooth/teeth. The best clinical gain is the minimal tooth preparation or no need for the removal of tooth substance. Treatment for this type of bridges does not usually require anaesthesia. In addition, adhesive bridges can provide reasonable aesthetical outcome with minimal cost and reduced chair time.

The biggest issue is that high failure rate in the long term, and gray colour shining through the metal wing cemented onto the abutment tooth. This can compromise the aesthetical outcome. The aesthetical problem can be solved by the use of zirconia all ceramic material to construct the bridge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Has a maximum of 2 units requiring placement
* Is a regular dental attendee and agree to return for assessments
* Written subject informed consent (IC) for this protocol will be obtained prior to study enrolment. Each subject will be required to sign and date the IC form prior to their participation
* Sound or minimally restored abutment(s)

Exclusion Criteria:

* The presence of any periodontal pocket depths equal or above 4 mm with active periodontal disease
* Any history of adverse reaction to clinical materials to be used in this study
* They are pregnant or had serious medical condition that may interfere with the dental treatment
* Acquired tooth loss more than 2 units requiring replacement
* Participants who have parafunctional habits
* Severe Class II Div II cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Clinical survival of adhesive bridges | 5 Years
  Evaluation of clinical survival: participants will be evaluated according to the modified USPHS criteria. The evaluation criteria will include: retention, framework fracture, veneering fracture, marginal adaptation, recurrent caries and colour match. The examination will be after one to two weeks, after 3, 6, 9, 12 and 18 months, 2, 3, 4 and 5 years. The evaluation will also include the biological complication. Plaque, gingival index, periodontal probing depth and gingival recession will be evaluated around the abutments and compared to a control tooth

SECONDARY OUTCOMES:
Quality of life, aesthetic outcome. | 18 months
  The patients will be requested to fill the OHIP-14 and the VAS questionnaires after one week to two weeks, after 3, 6, 9, 12 and 18 months in order to assess the quality of their lives and their aesthetic outcome after having the bridge.
Marginal discrepancy evaluation. | After cementation
  Marginal discrepancy will be evaluated by means of Scannining Electron Microscope (SEM) after cementation.
Economic evaluation | 5 years
  Economic evaluation will be run in parallel to the study and will include the overall cost of the two treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Baysan, BDS, MSc, PhD, Principal Investigator — Queen Mary University of London; Amani Agha, BDS,MSc, Study Director — Queen Mary University of London
Locations (1):
- Barts and The London, School of Medicine and Dentistry, London, United Kingdom